CLINICAL TRIAL: NCT06799013
Title: A Phase 1, Open Label, Dose-Escalation Study to Evaluate the Safety, Reactogenicity and Immunogenicity of a Nanoparticle Carrier-Formulated Self-Amplifying RNA Vaccine Against Crimean-Congo Hemorrhagic Fever (HDT-321) in Healthy Adults
Brief Title: Safety and Immunogenicity of a Self-Amplifying RNA Vaccine Against Crimean-Congo Hemorrhagic Fever
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HDT Bio (Industry)
Collaborators: DFNet Research Inc. (Other); Technical Resources International, Inc. (TRI) (Unknown); BioAgilytix Labs, LLC (Unknown); The University of Texas Medical Branch, Galveston (Other); Clinical Trials of Texas, Inc. (Other); Quest Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HDT-321-001; W15QKN-16-9-1002 / 23-86397-01 (Other Grant/Funding Number: Medical CBRN Defense Consortium (MCDC))
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Vaccine; Crimean-Congo Hemorrhagic Fever
Keywords: Vaccine; Healthy; 18-64; Male; Female; Preventative
MeSH Terms: conditions — Hemorrhagic Fever, Crimean

STUDY DESIGN:
Intervention Model Description: Four groups of 12 participants across three dose levels will be sequentially recruited in the study, starting with the lowest dose. The three dose levels and four treatment groups are outlined below.
  Group 1: 12 participants receive 10 μg vaccinations on Day 1 and Day 29 Group 2: 12 participants receive 25 μg vaccinations on Day 1 and Day 29 Group 3: 12 participants receive 50 μg vaccination on Day 1 Group 4: 12 participants receive 50 μg vaccinations on Day 1 and Day 29
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Group 1 will include 12 participants who will receive a 10 ug two dose schedule of HDT-321 at day 1 and day 29.
  Interventions: Biological: 10 ug HDT 321
- Group 2 (Experimental): Group 2 will include 12 participants who will receive a 25 ug, two dose schedule of HDT-321 at day 1 and day 29.
  Interventions: Biological: 25ug HDT-321
- Group 3 (Experimental): Group 3 will include 12 participants who will receive a 50 ug one dose schedule of HDT-321 at day 1.
  Interventions: Biological: 50ug HDT-321
- Group 4 (Experimental): Group 4 will include 12 participants who will receive a 50 ug two dose schedule of HDT-321 at day 1 and day 29.
  Interventions: Biological: 50ug HDT-321

INTERVENTIONS:
Biological: 10 ug HDT 321 — HDT-321 Investigational Vaccine (a Nanoparticle Carrier-Formulated self-amplifying RNA encoding the NP of CCHFV)
  Arms: Group 1
Biological: 25ug HDT-321 — HDT-321 Investigational Vaccine (a Nanoparticle Carrier-Formulated self-amplifying RNA encoding the NP of CCHFV)
  Arms: Group 2
Biological: 50ug HDT-321 — HDT-321 Investigational Vaccine (a Nanoparticle Carrier-Formulated self-amplifying RNA encoding the NP of CCHFV)
  Arms: Group 3; Group 4

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability and immunogenicity of three dosage levels, and a single or two-dose administration regimen, of the investigational HDT-321 product administered intra-muscularly. The main questions it aims to answer are:

* Is HDT-321 safe to use
* Does HDT-321 provide protection against Crimean-Congo hemorrhagic fever virus (CCHFV)

Researchers will record any adverse events and test blood samples to see if HDT-321 is safe and works to protect participants against Crimean-Congo hemorrhagic fever virus (CCHFV)

Participants will:

* Receive 1 or 2 doses of HDT-321
* Complete a memory aid and measurements for 7 days after receiving each dose of HDT-321
* Be followed throughout the study using phone calls and clinic visits to check for and record adverse events
* Provide blood samples at specific study visits

DETAILED DESCRIPTION:
This is an open-label, dose-escalation, first-in-human study to evaluate the safety, reactogenicity and immunogenicity of the investigational product HDT-321 in approximately 48 healthy adults aged 18-64 years.

Four groups of 12 participants at three dosage levels will be sequentially recruited in the study, starting with the lowest dose. Groups 1, 2 and 4 will receive 2 doses and group 3 will receive 1 dose of HDT-321.

Study progression and dose escalation will occur according to the following:

Group 1 (10 μg): Three sentinel participants will be initially enrolled and followed for 7 days post-first study injection for safety assessment by predetermined objective criteria. If none of the pre-defined halting rules are met, as confirmed by the Safety Review Team (SRT), enrollment of the remaining participants of the group will proceed. In addition, available safety data for 7 days post-second study injection will be evaluated in the sentinel group prior to administering the second injection of the remaining participants of Group 1. Available safety data for 7 days post-first study injection of all participants will be reviewed by the SRT. If none of the pre-defined halting rules are met and no safety concerns have been identified, enrollment of Group 2 participants will proceed.

Group 2 (25 μg): In a similar fashion, three sentinel participants will be initially enrolled and followed for 7 days post-first study injection for safety assessment by predetermined objective criteria. If none of the pre-defined halting rules are met, as confirmed by the SRT, enrollment of the remaining participants of the group will proceed. In addition, available safety data for 7 days post second study injection will be evaluated in the sentinel group prior to administering the second injection of the remaining participants of Group 2. Available safety data for 7 days post-first study injection of all Group 1 and 2 participants along with any available post-second injection from Group 1 participants will be reviewed by the SRT. If none of the pre-defined halting rules are met and no safety concerns have been identified, enrollment of Groups 3 and 4 participants will proceed.

Groups 3 and 4 (50 μg): the same procedure with initial enrollment of three sentinel participants will be followed as outlined above, prior to enrollment of the remaining participants of Group 3 and all of Group 4. In addition, the available data 7 days post-first injection of the entire Group 3 and 4 along with available post-second injection data from Group 1 and 2 will be reviewed prior to administering the second dose of Group 4 participants.

Blood samples will be collected from all participants in the study. Participants in groups 1, 2 and 4 will provide samples at screening and 8 additional visits. Participants in group 3 will provide samples at screening and 7 additional visits.

Participants will be requested to attend a combination of in person clinic visits and phone calls. Participants in groups 1, 2 and 4 will have 2 phone calls and 10 in-clinic visits. Two of the clinic visits will include administration of HDT-321 via IM injections. Participants in cohort 3 will have 1 phone call and 9 in-clinic visits. One of the clinic visits will include administration of HDT-321 via IM injection.

Protocol-defined solicited local and systemic AEs will be collected for 7 days following each study injection via memory aid. Other AEs will be collected for 28 days following each study injection. SAEs, AESIs, MAAEs and NOCDs will be collected from the first study injection through their entire study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females 18 to 64 years of age at the time of signing the ICF.
2. Body mass index (BMI) 17 to 35 inclusive at screening.
3. Considered by the PI or designee to be in good general health as determined by medical history, physical examination, vital sign measurements*, and clinical laboratory assessments conducted no more than 30 days prior to the first study injection administration.
4. Screening laboratory values within the laboratory reference ranges or considered non-clinically significant (NCS) if within Grade 1 severity on the toxicity grading scale.
5. Negative human immunodeficiency virus (HIV) 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
6. Women of childbearing potential must agree to use or have practiced true abstinence or use at least one acceptable primary form of contraception3 for at least 30 days prior to the first injection and for 60 days after the last injection. Female participants of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the day of and prior to each study injection.
7. Able to understand and comply with planned study procedures and willing to be available for all study required procedures, visits, and telephone calls for the duration of the study.
8. Provide written informed consent before initiation of any study procedures.
9. Willing to abstain from donating whole blood or blood derivatives 30 days prior to screening and for the duration of the study.
10. Willing to refrain from receiving any licensed vaccine within 28 days prior to and after scheduled study injections.

Exclusion Criteria:

1. Any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes study participation. Including Acute, subacute, intermittent, or chronic medical diseases or conditions that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of the trial. Significant respiratory disease (COPD) requiring daily medications, asthma that is not well controlled, significant cardiovascular disease, history of myocarditis or pericarditis, myocardial infarction, coronary artery bypass surgery or stent placement, or uncontrolled cardiac arrhythmia, Neurological or neurodevelopmental conditions, ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, blood dyscrasias or significant disorder of coagulation, chronic liver disease, including fatty liver, autoimmune disease, including localized or history of psoriasis or hypothyroidism without a defined non-autoimmune cause and Immunodeficiency of any cause.
2. Abnormal screening electrocardiogram (ECG)
3. History of hypersensitivity or severe reactions to previous vaccinations
4. History of hypersensitivity or severe reactions to products known to contain polyethylene glycol (PEG).
5. Allergy to antibiotics structurally similar to kanamycin (including but not limited to neomycin, streptomycin, tobramycin, and gentamycin).
6. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immunemodifying drugs within 6 months prior to the first study injection (for corticosteroids: prednisone ≥20 mg/day or equivalent). Intra-articular, inhaled, nasal, and topical steroids are allowed.
7. Received immunoglobulins or any blood products within 60 days prior to enrollment/Day 1.
8. Donated blood products within 30 days prior to enrollment/Day 1.
9. Received an investigational or non-registered medicinal product within 30 days prior to screening.
10. Currently enrolled, or plan to participate, in another clinical trial with an investigational agent to be received during the study period.
11. Received or plans to receive any non-study vaccine within 28 days before and after each study injection.
12. Febrile illness*, as determined by the participating site PI or appropriate sub-investigator, with or without fever (oral temperature ≥38.0°C/100.4°F), within 24 hours prior to each study injection.
13. Current heavy smoking/vaping (defined as 1 pack or more of cigarettes a day or vaping equivalent*). *1-2 mL of 20 mg/mL of nicotine salt
14. Known or suspected alcohol or illicit drug abuse within the past 12 months prior to Study Day 1.
15. Breastfeeding or plans to breastfeed from the time of the first vaccination through 60 days after the last study injection.
16. Participants unlikely to cooperate with the requirements of the study protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Solicited local and systemic adverse events (AEs) | Day 1-7 post administration
  Frequency and grade of solicited local and systemic AEs during the 7-day follow-up period after each study injection (i.e. the day of administration and 6 subsequent days).
Unsolicited study product related adverse events | Day 1-28 post administration
  Frequency and grade of unsolicited study product related AEs reported during the 28-day follow-up period after each study injection.
Laboratory abnormalities | Day 1-7 post administration
  Occurrence of laboratory abnormalities at 7 days post injection visit (increased or decreased outside normal ranges, as determined by the FDA Guidance for Industry Toxicity Grading Scale for Healthy Adults Enrolled in Preventive Vaccine Clinical Trials, 2007)
Serious AEs, AEs of Special Interest, Medically Attended AEs, and New-Onset of Chronic Diseases | Day 1 to end of study participation (Day 394)
  Frequency and grade of Serious AEs (SAEs), AEs of Special Interest (AESIs), Medically-Attended AEs (MAAEs), and New-Onset of Chronic Diseases (NOCDs) during the duration of participation in the study.

SECONDARY OUTCOMES:
Immunogenicity of HDT-321 | Day 1 to Day 57
  Evaluate the immunogenicity of HDT-321 as measured by IgG ELISA to the CCHFV NP measured 28 and 56 days after each injection. Using geometric mean titers (GMTs) of circulating antibodies against CCHFV NP through Day 57 along with seroconversion rate for anti-NP antibody through Day 57.

OTHER OUTCOMES:
Exploratory immunogenicity of HDT-321 | Day 1 to end of study participation (Day 394)
  Evaluate antibody subclass response as measured by IgG1, IgG2, IgG3, and IgG4 ELISA to the CCHFV NP. Using geometric mean titers (GMT) of antigen-specific IgG1, IgG2, IgG3, and IgG4.
Exploratory immunogenicity of HDT-321 | Day 57 to the end of study participation (Day 394)
  Evaluate the immunogenicity of HDT-321 as measured by IgG ELISA to the CCHFV NP measured after Day 57. Using geometric mean titers (GMTs) of circulating antibodies against CCHFV NP and seroconversion rate for anti-NP antibody.
Exploratory Immunogenicity of HDT-321 | Day 1 to end of study participation (Day 394)
  Evaluate the immunogenicity of HDT-321 vaccine as measured by IgG ELISA to the CCHFV NP from other strains. Using geometric mean titers (GMT) of strain-specific, antigen-specific IgG.
Exploratory immunogenicity of HDT-321 | Day 1 to end of study participation (Day 394)
  evaluate the immunogenicity as measured by IgM and IgA ELISA to the CCHFV NP. Using geometric mean titers (GMT) of antigen-specific IgM and IgA
Exploratory immunogenicity of HDT-321 | Day 1 to end of study participation (Day 394)
  evaluate B cell and T cell responses to CCHFV NP as percentages. Using the diversity of the cellular responses by assessing cells expressing interferon gamma (IFN-γ), interleukin 2 (IL-2), tumor necrosis factor (TNF), and other markers. as well as rate of antigen-specific cell-mediated immune responses for T cells expressing IFN-γ.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Duthie, PhD, Study Director — HDT Bio
Locations (1):
- Flourish Research San Antonio (Clinical Trials of Texas), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No